CLINICAL TRIAL: NCT04313803
Title: Expanding Continuous CGM Usage to Improve Outcomes in a Shorter Duration in Utah Valley Clinics
Brief Title: CGM in Utah Valley
Acronym: CGM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IHC IRB#: 1051315
Record Dates: First submitted 2020-03-13; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes
Keywords: Continuous glucose monitor (CGM); diabetes; glucose
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- American Fork: CGM usage months 1 and 3
  Interventions: Device: CGM
- Central Orem: CGM usage for month 1
  Interventions: Device: CGM
- North Canyon, Saratoga Springs, and Lehi: CGM usage for 1-3 months
  Interventions: Device: CGM

INTERVENTIONS:
Device: CGM — Dexcom CGM system

SUMMARY:
The purpose of this study is to replicate the positive impact observed in IRB #1050955, but conduct this over a shorter period to potentially maximize patient outcomes and make care more affordable. Intermountain intends to build a diabetes program with CGM based on the findings. Senior stakeholders, clinicians and operators are aligned on this vision including the Community Based Care triad, Executive Leadership Team, and our Diabetes Prevention Program.

DETAILED DESCRIPTION:
Overview

Approximately 30 million Americans, or 9% of the population has diabetes, a condition in which a person does not make enough insulin, or the body cannot use its own to effectively manage blood glucose levels. Improper diabetes management is associated with severe comorbidities which include: heart disease, stroke, kidney disease, ocular problems, dental disease, nerve damage, and vascularity issues. The epidemic continues to challenge systems like Intermountain Healthcare, an accountable care organization (ACO), since diabetes cost $327 billion per year (representing $1 in every $7 dollars spent) on healthcare in the United States. Furthermore, people with diagnosed diabetes incur average medical expenditures of $16,752 per year, of which about $9,601 is directly attributed to diabetes. New treatment options are needed to manage population health, especially with 84 million adults having been diagnosed with prediabetes diabetes.

In an effort to reduce the physical, economic and social burden of diabetes, several healthcare systems have evaluated the use of telehealth to monitor glucose levels. In a previous metanalysis, the authors demonstrated that telehealth interventions produced a small, but significant improvement in hemoglobin A1c (HbA1c) levels compared with usual care (mean difference: -0.55, 95% CI: -0.73 to - 0.36). The Ontario Health Technology Advisory Committee also showed that the blood glucose home telemonitoring technologies they used yielded a statistically significant reduction in HbA1c of ~0.50% in comparison to usual care when used adjunctively to a broader telemedicine initiative for adults with type 2 diabetes.

1.2 Previous Work

Intermountain Healthcare conducted a pilot study in the Reimagine Primary Care (RPC) clinics to evaluate if six months of CGM could improve patient outcomes (IRB #1050955). A total of 99 patients remained enrolled for the full time period (n=50 CGM, n=49 standard of care (SOC)), and data showed a improvement in glucose levels, less primary care and specialty appointments, a reduction in emergency department (ED) encounters, less labs ordered, and a cumulative body mass index (BMI) improvement. Furthermore, nearly all participants reported being willing to engage in another future pilot, and the vast improvements were attributed to subjects use of real-time data.

Primary analyses

Cost of care for fee-for-value patients (specifically PMPM savings)

Secondary analyses

Frequency of hypoglycemic events, healthcare utilization per count of inpatient/outpatient visits, cost of care, current HEDIS performance on diabetes and behavioral health measures, coding specificity for diabetes, emergency department visit per 1000 rate, overall and for patients with diabetes.

Power analyses

Data from IRB #1050955 has shown significant changes in cost, care and utilization with only a sample of 50 CGM users. The effect size is currently being calculated by the study statistician, but most of the outcome variables comparing CGM to standard of care device were p<0.05. Given that this will now include a much larger population, and 30x participant increase, the investigators will have sufficient power to deduce differences should they occur.

ELIGIBILITY:
Inclusion Criteria:

* Patients (18-80 years of age) with type ll diabetes, having an HbA1c ≥6.5%, treated within five Intermountain Healthcare Utah Valley clinics. Patients must have access to a smart phone to download applications, have Bluetooth capabilities for data sharing, and log/view their continuous glucose monitor (CGM) data.

Exclusion Criteria:

* Patients who are pregnant, not classified as having diabetes based on A1c levels, and age ≤ 17 or ≥ 81 years, or diagnosis of dementia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with type II diabetes treated at Intermountain Healthcare
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Cost of care for fee-for-value patients (specifically PMPM savings) | 1 April 2020 - 30 April 2021
  For each patient, measure total variable cost of associated healthcare services and visits. Then compare the distribution of costs between randomized groups using the Wilcoxon rank-sum test, a non-parametric analogue of Student's t-test.

SECONDARY OUTCOMES:
The count of primary care, specialist, and emergency department visits or hospital stays for those using CGM compared to historical utilization and the broader T2DM cohort within Intermountain Healthcare. | 1 April 2020 - 30 April 2021
  Frequency of hypoglycemic events and healthcare utilization per count of inpatient/outpatient and emergency department visits per 1000 rate, overall and for patients with diabetes
Evaluation of HEDIS performance for those using CGM compared to historical utilization and the broader T2DM cohort within Intermountain Healthcare. | 1 April 2020 - 30 April 2021
  Current HEDIS performance on diabetes and behavioral health measures

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Joy, MD, MPH, Principal Investigator — Intermountain Health Care, Inc.; Brad Isaacson, PhD, MBA, MSF, PMP, Study Director — Intermountain Health Care, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee PA, Greenfield G, Pappas Y. The impact of telehealth remote patient monitoring on glycemic control in type 2 diabetes: a systematic review and meta-analysis of systematic reviews of randomised controlled trials. BMC Health Serv Res. 2018 Jun 26;18(1):495. doi: 10.1186/s12913-018-3274-8. PMID 29940936
- [Background] Ekhlaspour L, Mondesir D, Lautsch N, Balliro C, Hillard M, Magyar K, Radocchia LG, Esmaeili A, Sinha M, Russell SJ. Comparative Accuracy of 17 Point-of-Care Glucose Meters. J Diabetes Sci Technol. 2017 May;11(3):558-566. doi: 10.1177/1932296816672237. Epub 2016 Oct 3. PMID 27697848
- [Background] Verkuilen J. Explanatory Item Response Models: A Generalized Linear and Nonlinear Approach by P. de Boeck and M. Wilson and Generalized Latent Variable Modeling: Multilevel, Longitudinal and Structural Equation Models by A. Skrondal and S. Rabe-Hesketh. Psychometrika. 2006 Jun;71(2):415-418. doi: 10.1007/s11336-005-1333-7. No abstract available. PMID 28197954
- [Background] Fong Y, Rue H, Wakefield J. Bayesian inference for generalized linear mixed models. Biostatistics. 2010 Jul;11(3):397-412. doi: 10.1093/biostatistics/kxp053. Epub 2009 Dec 4. PMID 19966070